CLINICAL TRIAL: NCT01278134
Title: INFORM-SVR: A Randomized, Multi-Center Study of Interferon-Free Treatment With a Combination of a Polymerase Inhibitor (RO5024048) and a Ritonavir Boosted HCV Protease Inhibitor (RO5190591/r, DNV/r) With or Without Copegus® in Interferon Naïve HCV Genotype 1 Infected Patients
Brief Title: A Study of RO5024048 in Combination With Ritonavir-Boosted Danoprevir With or Without Copegus (Ribavirin) in Interferon-Naïve Patients With Chronic Hepatitis C Genotype 1 (INFORM-SVR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP25213; 2010-022067-35
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — danoprevir; peginterferon alfa-2a; Ribavirin; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm B Extension (Experimental): All patients in treatment arm B were offered to receive Pegasys/Cogepus therapy for an additional 24 weeks.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]
- RO5024048 & ritonavir-boosted danoprevir without Ribavirin (B) (Experimental)
  Interventions: Drug: Copegus placebo; Drug: RO5024048; Drug: danoprevir; Drug: ritonavir
- RO5024048 and ritonavir-boosted danoprevir with Ribavirin (A) (Experimental)
  Interventions: Drug: RO5024048; Drug: danoprevir; Drug: ribavirin [Copegus]; Drug: ritonavir

INTERVENTIONS:
Drug: Copegus placebo — 1000 mg or 1200 mg daily orally in split doses (morning/evening), up to 24 weeks
  Arms: RO5024048 & ritonavir-boosted danoprevir without Ribavirin (B)
Drug: RO5024048 — 1000 mg bid orally, up to 24 weeks
  Arms: RO5024048 & ritonavir-boosted danoprevir without Ribavirin (B); RO5024048 and ritonavir-boosted danoprevir with Ribavirin (A)
Drug: danoprevir — 100 mg bid orally, up to 24 weeks
  Arms: RO5024048 & ritonavir-boosted danoprevir without Ribavirin (B); RO5024048 and ritonavir-boosted danoprevir with Ribavirin (A)
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly, 24 weeks
  Arms: Arm B Extension
Drug: ribavirin [Copegus] — 1000 mg or 1200 mg daily orally in split doses (morning/evening), up to 24 weeks
  Arms: Arm B Extension; RO5024048 and ritonavir-boosted danoprevir with Ribavirin (A)
Drug: ritonavir — 100 mg bid orally, up to 24 weeks
  Arms: RO5024048 & ritonavir-boosted danoprevir without Ribavirin (B); RO5024048 and ritonavir-boosted danoprevir with Ribavirin (A)

SUMMARY:
This multicenter, randomized, double-blind, parallel group study will evaluate the safety and efficacy of the combination RO5024048 and ritonavir-boosted danoprevir with and without Copegus (ribavirin) in patients with chronic hepatitis C genotype 1. In arm A and B, interferon treatment-naïve patients will receive 1000 mg RO5024048 orally twice daily and 100 mg danoprevir with 100 mg ritonavir orally twice daily plus either Copegus (1000 mg or 1200 mg orally daily) or placebo for 12 weeks. Depending on viral response and treatment arm patients will be re-randomized to continue assigned treatment for additional 12 weeks or stop all treatment. The anticipated time on study treatment is up to 24 weeks plus a 24-week follow-up.

As of 29. September 2011, Arm B patients (placebo-containing arm) will be offered, in conjunction with the current treatment, Pegasys (peginterferon alfa-2a) 180 mcg subcutaneously weekly plus Copegus 1000mg or 1200 mg orally daily for 24 weeks, with a 24-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, >/= 18 years of age
* Chronic Hepatitis C of >/= 6 months duration at screening
* HCV genotype 1 and quantifiable HCV RNA at screening (Roche COBAS TaqMan HCV test)
* Naïve for treatment with interferon (pegylated or non-pegylated)
* Body Mass Index (BMI) 18-35 inclusive, minimum weight 45 kg
* Females of child-bearing potential and males with female partners of childbearing potential must use 2 forms of effective non-hormonal contraception

Exclusion Criteria:

* Pregnant or lactating women and males with female partners who are pregnant or lactating
* Decompensated liver disease or impaired liver function
* Cirrhosis or incomplete/transition to cirrhosis
* Non-hepatitis C chronic liver disease
* Hepatitis B or HIV infection
* History of neoplastic disease within the last 5 years, except for localized or in situ carcinoma of the skin
* History of pre-existing renal disease (except for nephrolithiasis) or severe cardiac disease
* History of drug or alcohol abuse within the last year or alcohol consumption of > 2 units per day; cannabinoid use is excepted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Sustained virological response, defined as undetectable HVC RNA measured by Roche COBAS TaqMan HCV test | 24 weeks after end of treatment
Safety: Incidence of adverse events | 1.5 years

SECONDARY OUTCOMES:
Virological response (HCV RNA measured by Roche COBAS Taqman HCV test) | up to 48 weeks
Impact of Copegus (ribavirin) on efficacy of the direct-acting antiviral combination regimen: viral response (HCV RNA measured by Roche COBAS TaqMan HCV test) | 1.5 years
Comparison of 12 and 24 weeks of treatment duration: viral response (HCV RNA measured by Roche COBAS TaqMan HCV test) | 1.5 years
Pharmacokinetics: Plasma concentrations of danoprevir, ritonavir, RO4995855 (parent drug of RO5024048) and ribavirin | up to 24 weeks
Viral resistance: HCV RNA sequencing and phenotypic analyses | up to 48 weeks
Effect of interleukin 28B genotype on efficacy: viral response (HCV RNA measured by Roche COBAS TaqMan HCV test) | 1.5 years
Quality of life: SF-36 questionnaire, Fatigue Severity Scale | up to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (17):
  - La Jolla, California
  - Sacramento, California
  - Orlando, Florida
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lutherville, Maryland
  - Detroit, Michigan
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Houston, Texas
  - Newport News, Virginia
  - Vancouver, Washington
- France (6):
  - Clichy
  - Créteil
  - Lille
  - Marseille
  - Montpellier
  - Paris
- Germany (6):
  - Berlin
  - Frankfurt am Main
  - Hamburg
  - Hanover
  - Kiel
  - Leipzig
- Grafton, New Zealand

REFERENCES:
- [Derived] Tong X, Li L, Haines K, Najera I. Identification of the NS5B S282T resistant variant and two novel amino acid substitutions that affect replication capacity in hepatitis C virus-infected patients treated with mericitabine and danoprevir. Antimicrob Agents Chemother. 2014 Jun;58(6):3105-14. doi: 10.1128/AAC.02672-13. Epub 2014 Mar 17. PMID 24637689